CLINICAL TRIAL: NCT04858282
Title: Department of Nursing, Chang Gung Memorial Hospital-Kaohsiung Medical Center,RN, MSN
Brief Title: Application-Enabled Shared Decision-Making
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chia-Wen,Chuang, Department of Nursing, RN, MSN, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: mavis20023
Record Dates: First submitted 2021-04-16; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Mastectomy; Breast-Conserving Surgery
Keywords: early breast cancer; surgery; shared decision-making; m-health; application; patient decision aid
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- shared decision-making group (SDMG) (Experimental): Receiving mobile application( BC-SDM)
  Interventions: Other: mobile application (BC-SDM)
- usual care group (UCG) (No Intervention): Receiving material health education

INTERVENTIONS:
Other: mobile application (BC-SDM) — The mobile application (BC-SDM)includes four functions to support SDM activity: "Understanding breast cancer," "Surgical approach," "Choose the right breast cancer knowledge," and "Let's make a decision for myself". Patients first read the information in "Understanding breast cancer" and "Surgical approach" to receive a tailored education in breast cancer
  Arms: shared decision-making group (SDMG)

SUMMARY:
To develop application-enabled shared decision-making among patients with early breast cancer and evaluate the preliminary effects of the interventions.

DETAILED DESCRIPTION:
Female breast is an amazing organ that it symbolizes not only the female gender, but also the continuity of human race. In the past treating breast cancer may signal a termination of the breast's predestined role in a woman or a mother. Nowadays, surgical treatment of early breast cancer has two options, one is breast-conserving surgery and the other one is total mastectomy. The former treatment option preserves most of the breast tissue but may spare dormant cancer cells in the preserved tissue. The latter treatment option spares no breast tissue and as a result no dormant cancer cells would remain. This treatment dilemma may bother most of the patients especially when they are still under the shade of the bad news. Many women are reluctant to discuss their diseased breasts with their folks or even their doctors because of privacy; instead they would seek information through internet. Unfortunately, most of their final decision is doctor's preferred choice despite they may have doubts or concerns on doctor's choice of treatment.

Share decision making (SDM) is a recently developed strategy that allows patients taking part in their treatment plan. Patients are invited to join the meeting where doctors explain the latest treatment options and patients express their concerns and finally a decision, both doctors' and patients' concerns well integrated, is reached. One of the drawbacks of SDM is too time consuming; doctors have to prepare a lot of pertinent information, while patients have to try their best to understand the provided information, though many patients may not fully understand their treatment options. It has been reported that a well designed patient decision aids (PDAs) could serve as a virtue connection between patients and doctors. Instead of merely taking information from the PDAs, it allows patients to know all the possible options of treatment and the side effects in an interactive way. It is supposed that patients could be well prepared to discuss with their doctors after interaction with the customized PDAs. In Taiwan, decision conflict and decision regret are commonly encountered among most cancer patients. The impetus for developing a PDAs for female breast cancer patients and evaluating its role on lowering decision conflict and decision regret among these patients comes from the high rates of decision conflict and decision regret among cancer patients in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* women, aged >20 years
* newly diagnosed early breast cancer (stages 0-II)
* no surgery yet
* no metastases
* tumor size <3 cm

Exclusion Criteria:

•tumor located <2 cm from the nipple

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
knowledge tests | immediately after the intervention
  The knowledge tests included five items,1. Are the survival rates of breast cancer the same with conserving surgery and total mastectomy? 2. Breast-conserving surgery has a higher local-regional recurrence rate? 3. Is radiation therapy required for Breast-conserving surgery? 4. Does total mastectomy require longer recovery time? 5. Do both total mastectomy and breast-conserving surgery have the same bleeding and infection rate? The knowledge tests included five items, such as "Are the survival rates of breast cancer the same with conserving surgery and total mastectomy?" The correct answer was coded as one point. The scores of the knowledge tests ranged from zero to five points. Higher scores indicated more correct knowledge.
decision conflict-sure | immediately after the intervention
  The Decision Conflict Scale (DCS_SURE) included four items: uncertainty, information, values clarity, and support and effective decision. On the scale, "Yes" answers scored one point, while "No" responses were zero points. The higher score, the lesser conflict.
Decision Regret Scale DRS | immediately after the intervention
  The Decision Regret Scale was composed of five items: "It was the right decision," "I regret the choice that was made," "I would go for the same choices if I had to do it over again," "The choices did me a lot of harm," and "The decision was a wise one." Items were scored using a five-point Likert scale, ranging from very agreed (1 point) to very disagreed (5 points), but two items were reversely scored. The higher score, the more regret.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No